CLINICAL TRIAL: NCT01671436
Title: Central Meditation and Imagery Therapy for Depression
Brief Title: Meditation for Depression
Acronym: CMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMIT-1042
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Depression
Keywords: Depression; Guided Imagery; Psychotherapy; Meditation
MeSH Terms: conditions — Depression | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Central Meditation and Imagery Therapy (Experimental): Intervention involved Central Meditation, may be characterized by a voluntary, regulated attentional set towards a specific stimulus or set of stimuli and visualization exercises utilized within CMIT, which primarily involves two types of thought experiments: 1) creating mental models of how a person fits into the larger world and universe according to evolutionary biology and modern cosmology, in order to gain a larger perspective on emotions and thought patterns, and 2) backcasting, the generation of a desirable future coupled with mental time travel back to the present to determine how to create that future with present-day actions.
  Interventions: Behavioral: Central Meditation and Imagery Therapy

INTERVENTIONS:
Behavioral: Central Meditation and Imagery Therapy

SUMMARY:
Major Depressive Disorder (MDD) is a serious, costly and highly prevalent condition. However, currently available treatment options have limited efficacy. The aim of this pilot study is to determine whether patients suffering from MDD who have not responded to at least one antidepressant trial may actively engage in a novel group therapy, Central Meditation and Imagery Therapy (CMIT). Preliminary results with individual patients suggest that CMIT techniques may have benefit for major depression. The purpose of this trial is to assess the feasibility of a group form of CMIT for the treatment of major depression. The trial will also seek to identify neurophysiological and cardiovascular predictors of treatment response.

In this study, 10 subjects with major depressive disorder will receive antidepressant treatment augmentation with group meditation and mental imagery therapy for a total of 12 weeks, as well as daily meditation practice. Group sessions will also involve gentle yogic stretches. The subjects will be limited to those who remain depressed despite at least one trial of antidepressant medication. Changes in brain activity and heart rate variability will be measured at three time points utilizing electroencephalography (EEG) and pulse monitors. Depression symptoms will be measured at several time points using questionnaires and objective measures. Participation will require a total of 15 visits for weekly therapy and the measurements. Two-month follow-up questionnaires will be mailed to the subjects after study end to assess durability of any improvements in depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the DSM-IV criteria for unipolar major depressive disorder, as assessed by the Mini-Neuropsychiatric International Interview (MINI).
* HAM-D17 rating scale ≥ 14.
* Prior treatment with antidepressant medication during the present major depressive episode
* Adequate written and oral fluency in English to understand and complete study forms and converse with study personnel.
* Willingness on part of both subject and treating clinician to not change antidepressant treatment, including medications, psychotherapy or other treatments, over the course of the study, unless necessary to provide for well being of subject.

Exclusion Criteria:

* Current diagnosis of schizophrenia or any psychotic disorder including psychotic depression, dysthymia, mania or bipolar disorder, attention deficit or hyperactivity disorder, generalized anxiety disorder or panic disorder, obsessive compulsive disorder, alcohol or drug dependence, mental retardation, any pervasive developmental disorder or cognitive disorder (according to DSM-IV) criteria. Those with lifetime history of psychiatric conditions other than unipolar major depression will be also excluded.
* Medically unstable, delirious, or terminally ill (e.g. medical illness requiring hospitalization or intense outpatient management, such as heart disease; heart attack in the past 6 months; congestive heart failure; severe heart arrythmias; unstable hypertension; poorly controlled diabetes; or pending surgery).
* Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke/ aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.
* Participants regularly practicing (≥ 2 times per week) any of the techniques utilized in the study to reduce stress: meditation, guided imagery, yoga.
* Current treatment with behavior therapy or psychotherapy.
* Active suicidal plan as measured by HAM-D item 3 score of greater than or equal to 3, or history of suicide attempt during the current episode.
* Utilization of cannabis or other illicit drugs more than once a month.
* Excessive use of alcohol, i.e., men whose alcohol consumption exceeds 14 standard drinks per week or 4 drinks per day, and women whose alcohol consumption exceeds 7 standard drinks per week or 3 drinks per day.
* Needing to adjust or change anti-depressant treatment, including medications, psychotherapy, repetitive Transcranial Magnetic Stimulation (rTMS), Electroconvulsive Therapy (ECT), or Vagus Nerve Stimulation (VNS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | Measured 4 times over 12 weeks
  Primary outcome is change in HAM-D from baseline to Week 12.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms- Self Report (QIDS- SR) | Weekly assessments measured over 12 weeks, and 2 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Jain, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States